CLINICAL TRIAL: NCT00899431
Title: Nonmyeloablative Stem Cell Transplantation With or Without Lenalidomide for Chronic Lymphocytic Leukemia (RV-CLL-PI-0294)
Brief Title: Nonmyeloablative Stem Cell Transplantation for Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated per PI's request at the time of continuing review
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0871; NCI-2012-01620 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Nonmyeloablative Stem Cell Transplantation; Chronic Lymphocytic Leukemia; CLL; Immunomanipulation; Fludarabine; Lenalidomide; Rituximab; Thymoglobulin; Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; fludarabine; fludarabine phosphate; Rituximab; thymoglobulin; Antilymphocyte Serum; Stem Cell Transplantation; Bendamustine Hydrochloride; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Lenalidomide (Active Comparator): Chemotherapy, Plus Lenalidomide - Lenalidomide starting dose 5 mg by mouth every other day; increase to 5 mg/d daily in 4-5 weeks for 6 - 12 months. Fludarabine 30 mg/m^2 intravenously daily on days -5, -4, -3. Rituximab 375 mg/m2 intravenously on day -13, and 1000 mg/m^2 on days -6, +1 and +8. Thymoglobulin 1.0 mg/kg intravenously over 4 hours (day -2 and -1). On Day 0, donor blood stem cells collected will be transplanted over 30-45 minutes. Bendamustine 130 mg/m2/day by vein daily on day -5, -4, -3 (following Fludarabine). Allopurinol 300 mg by mouth daily beginning at the start of lenalidomide therapy and continuing for 3 months.
  Interventions: Drug: Lenalidomide; Drug: Fludarabine; Drug: Rituximab; Drug: Thymoglobulin; Procedure: Stem Cell Transplantation; Drug: Bendamustine; Drug: Allopurinol
- Group 2: No Lenalidomide (Active Comparator): Chemotherapy Treatment, No Lenalidomide - Fludarabine 30 mg/m^2 intravenously daily on days -5, -4, -3. Rituximab 375 mg/m2 intravenously on day -13, and 1000 mg/m^2 on days -6, +1 and +8. Thymoglobulin 1.0 mg/kg intravenously over 4 hours (day -2 and -1). On Day 0, donor blood stem cells collected will be transplanted over 30-45 minutes. Bendamustine 130 mg/m2/day by vein daily on day -5, -4, -3 (following Fludarabine).
  Interventions: Drug: Fludarabine; Drug: Rituximab; Drug: Thymoglobulin; Procedure: Stem Cell Transplantation; Drug: Bendamustine

INTERVENTIONS:
Drug: Lenalidomide — Starting dose 5 mg by mouth every other day; increase to 5 mg/d daily in 4-5 weeks for 6 - 12 months
  Other Names: CC-5013; Revlimid
  Arms: Group 1: Lenalidomide
Drug: Fludarabine — 30 mg/m^2 intravenously daily on days -5, -4, -3.
  Other Names: Fludara; Fludarabine Phosphate
Drug: Rituximab — 375 mg/m2 intravenously on day -13, and 1000 mg/m^2 on days -6, +1 and +8.
  Other Names: Rituxan
Drug: Thymoglobulin — 1.0 mg/kg intravenously over 4 hours (day -2 and -1).
  Other Names: ATG; rabbit anti-thymocyte globulin
Procedure: Stem Cell Transplantation — On Day 0, donor blood stem cells collected will be transplanted over 30-45 minutes.
  Other Names: SCT; Nonmyeloablative Stem Cell Transplantation
Drug: Bendamustine — 130 mg/m2/day by vein daily on day -5, -4, -3 (following Fludarabine).
  Other Names: Bendamustine Hydrochloride; Bendamustine HCL; CEP-18083; SDX-105; Treanda
Drug: Allopurinol — 300 mg by mouth daily beginning at the start of lenalidomide therapy and continuing for 3 months.
  Other Names: Lopurin; Zurinol; Zyloprim
  Arms: Group 1: Lenalidomide

SUMMARY:
The goal of this clinical research study is to learn if lenalidomide, when given with a stem cell transplant and chemotherapy (bendamustine, fludarabine, and rituximab), can help to control CLL. The safety of this treatment combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

Bendamustine is designed to damage and destroy the DNA (genetic material) of cancer cells.

Fludarabine is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells). This may increase the likelihood of the cells dying.

Rituximab is designed to attach to leukemia cells, which may cause them to die.

Before receiving the study drugs, 21 or more days must have passed since your last biological therapy, chemotherapy, radiotherapy, or other investigational therapy.

Before you begin therapy, you will have the following tests and procedures performed. The blood may need to be drawn daily. The doctor will tell you how often the other tests will need to be performed:

* You will have a physical exam.
* You will have blood transfusions of blood and platelets as needed.
* Blood (about 2 tablespoons) and urine will be collected for routine tests.
* Blood (about 6-10 tablespoons) will be drawn to check the effects of the transplant.
* You will have a chest x-ray and CT scans to check the status of the disease.
* You will have an ECG.
* You will have a bone marrow biopsy and aspirate, when the doctor thinks it is needed.

Study Treatment:

If you are found to be eligible to take part in this study, you will begin treatment within 30 days after the screening visit. All liquid study drugs will be given through a central venous catheter (CVC) that will be left in place throughout treatment. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

On Days -13, -6, +1, and +8, you will receive rituximab over 5-7 hours by CVC.

On Days -5 to -3, you will receive fludarabine over 1 hour and bendamustine over 1 hour by CVC. You will be given standard drugs such as hydrocortisone and Tylenol to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

On Days -2 to -1, if the donor is not related or is not completely matched, you will receive thymoglobulin (ATG) over 4 hours by CVC. This will help to reduce the risk of your body rejecting the transplant.

On Days -2 to -1, if the donor is related, you will "rest" (not receive chemotherapy).

On Day -2, you will start to receive tacrolimus by CVC to help prevent graft-versus-host disease. This will be changed to a dose of tacrolimus by mouth, once you are discharged from the hospital. You will continue to take tacrolimus by mouth for 6-8 months following your transplant.

On Day 0, the blood stem cells that were collected from your donor will be transplanted (given back to your body) through the CVC over 30-45 minutes.

On Days 1, 3, and 6 after the stem cell transplant (and Day 11 if the donor is not related or not completely matched), you will receive methotrexate over 30-60 minutes by CVC to help prevent graft-versus-host disease.

On Day 7 after the transplant, G-CSF (filgrastim) will be injected under your skin once a day until your white blood cell counts recover. Filgrastim is designed to help increase the number of white blood cells.

Treatment with Lenalidomide:

If your blood cell counts are high enough and if you have not experienced side effects, between Days 90 and 100 after the transplant, you will be randomly assigned (as in the flip of a coin) into 1 of 2 groups. If you are in Group 1 you will take lenalidomide in addition to the treatment listed above. If you are in Group 2, you will not take lenalidomide.

If you are in Group 1, you will take lenalidomide 1 time every day for 3-12 months, depending on the disease response to the treatment.

You should swallow lenalidomide capsules whole, with water, at the same time each day. Do not break, chew, or open the capsules.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

If you take more than the prescribed dose of lenalidomide you should seek emergency medical care (if needed) and contact the study staff right away.

You will be given standard drugs such as aspirin, Coumadin (warfarin), heparin, and/or allopurinol to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

If the doctor thinks it is needed, your dose and schedule of lenalidomide will be changed.

If you are in Group 2, you will take no additional drugs.

Pregnancy Tests While Taking Lenalidomide:

Women who are able to become pregnant must have 2 negative pregnancy tests: the first test within 10-14 days before lenalidomide is prescribed and the second test within 24 hours before lenalidomide is prescribed. This blood test will be taken as part of a routine blood draw. The prescription must be filled within 7 days.

Once a week for the first month you take lenalidomide, women who are able to become pregnant will have blood (about 1 teaspoon) drawn for a pregnancy test. Then, in females with regular menstrual cycles, blood (about 1 teaspoon) will be drawn for pregnancy testing every 4 weeks, at the end of study, and 28 days after the last dose of lenalidomide. If menstrual cycles are irregular, blood (about 1 teaspoon) will be drawn every 2 weeks, at the end of study, and 14 and 28 days after the last dose of lenalidomide.

Study Visits (both Groups):

You must stay in the Houston area for about 100 days after the stem cell transplant.

Between Days 25 and 35 and then about 3 months after the stem cell transplant:

* You will have a physical exam.
* You will have CT scans to check the status of the disease.
* You will have PET scan to check the status of the disease, if the doctor thinks it is needed.
* Blood (about 2 tablespoons) will be drawn for routine tests and to check the level of tacrolimus.
* You will have a bone marrow biopsy/aspirate to check the status of the disease.

Study Visits (Group 1):

If you are in Group 1, blood (about 2 tablespoons) will be drawn for routine tests weekly until the maximum dose of lenalidomide is reached, then once every 2 weeks while you are taking lenalidomide.

Follow-up:

Every 3 months during the first 18 months and then every 6 months up to 3 years:

* You will have a physical exam.
* You will have CT scans to check the status of the disease.
* You will have PET scans to check the status of the disease, if the doctor thinks it is needed.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a bone marrow biopsy to check the status of the disease.

Length of Study:

You will be on study up to about 3 years. You will be taken off study if the disease gets worse or you experience any intolerable side effects.

End-of-Study Visit:

After you are off study, you will have an end-of-study visit:

* You will have a physical exam.
* You will have CT scans to check the status of the disease.
* You will have PET scans to check the status of the disease, if the doctor thinks it is needed.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a bone marrow biopsy to check the status of the disease.

Data Confidentiality Plan:

Data will be collected in the SCT&CT departmental database (BMTWeb). This database is password-protected, contains audit tracking, and follows all federal guidelines. Your personal identifying information will be removed for this analysis; no sensitive information will be shared.

This is an investigational study. All of the drugs used in this study are FDA approved and commercially available for the treatment of CLL. The use of the drugs together in this study is investigational.

Up to 80 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years at the time of signing the informed consent form.
2. Disease: CLL in relapse, after failing conventional chemo-antibody combination therapy; CLL patients who failed to achieve CR with frontline conventional chemo-antibody; CLL patients with 17p deletion; CLL in Richter's.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Donor: HLA compatible related (HLA-A,-B,-DRBI matched or with one-antigen mismatched) or HLA compatible unrelated.
5. ECOG performance status of </= 2 at study entry
6. FEV1, FVC and DLCO >/= 40%.
7. Left ventricular EF > 40% with no uncontrolled arrhythmias or symptomatic heart disease.
8. Serum creatinine </= 1.6 mg/dL. Serum bilirubin < 1.6 mg/dL.
9. SGPT < 2x upper limit of normal.
10. Voluntary signed, written IRB-approved informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
11. All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 3 weeks prior to treatment in this study.
12. Disease free of prior malignancies for >/= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
13. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to study entry.
14. Disease must be chemosensitive (ie, patients must have PR or better based on CT Scans, PET Scan, and bone marrow biopsy).
15. Patients suspected to have Richter's transformation (such as elevated LDH) and/or who are PET positive, should have a lymph node biopsy to assess histological status of the disease
16. Patients must be off of alemtuzumab for 6 weeks prior to consenting.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide, lenalidomide, bendamustine, fludarabine. For patients will unrelated donors: Known hypersensitivity to thymoglobulin.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Concurrent use of other anti-cancer agents or treatments.
8. Known positive for HIV or infectious hepatitis, type A, B or C.
9. Sinuses should be evaluated by either CT neck or CT sinuses to exclude infections
10. Deep-vein thrombosis or pulmonary embolism within 3 months of study entry.
11. History of serious infection requiring hospitalization within the last 3 months of consenting.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-05-06 (Actual); Primary Completion 2018-10-07 (Actual); Study Completion 2018-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, BS, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from May 2009 to November 2012 for subjects with chronic lymphocytic leukemia (CLL) who had relapsed after failing conventional chemo-antibody combination therapy, or failed to achieve a Crwith frontline conventional chemo-antibody, or have 17p deletion, or in Richter's.
Pre-assignment Details: Patients were randomized at a 1:1 ratio to receive lenalidomide 90 to 100 days after allo SCT if they had persistent active CLL
Groups:
- Not Randomized: Did not meet the necessary criteria after transplantation to be randomized for maintenance.
- Randomized to Lenalidomide: 1:1 randomization. This group receive the study drug Lenalidomide.
- Randomized to Not Receive Lenalidomide: 1:1 randomized. This group did not receive lenalidomide.
Period: Overall Study
Arm/Group | Not Randomized | Randomized to Lenalidomide | Randomized to Not Receive Lenalidomide
Started | 22 | 8 | 9
Completed | 21 | 8 | 9
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Not Randomized
- Group 2: Randomized to Lenalidomide
- Group 3: Randomized to not receive lenalidomide
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 21 | 8 | 9 | 38
Age, Continuous [Median (Full Range); unit: Years] | 60 [45 to 72] | 55 [47 to 70] | 56 [45 to 72] | 58 [45 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 16 | 6 | 7 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 6
  White | 18 | 6 | 6 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 8 | 9 | 38
Conditioning regimen [Count of Participants; unit: Participants] — May 2009 to November February 2011 used the established regimen of Fludarabine-cyclophosphamide and rituximab (FCR). In August 2011 the conditioning regimen was changed to bendamustine, fludarabine, and rituximab (BFR).
  Participants
    FCR | 12 | 6 | 7 | 25
    BRF | 9 | 2 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Immunomanipulation After Non-myeloablative Stem Cell Transplantation for CLL (Chronic Lymphocytic Leukemia).
Description: To compare the need for immunomanipulation within 18 months after non-myeloablative allogeneic transplantation for CLL between the two combination therapies with or without lenalidomide maintenance. For this purpose, "immunomanipulation" is defined as any one of the following events: 1) Cessation of administering tacrolimus treatment with in the first 6 months after allotransplant due to persistent disease or progression. 2) Boost of donor lymphocytic infusion (DLI) administered anytime between 3 and 18 months after allotransplant.
Time Frame: Up to 18 months after allotransplant.
Population: Data were not collected due to low accrual of participants and protocol was terminated.
Arm/Group | Not Randomized | Randomized to Lenalidomide | Randomized to Not Receive Lenalidomide
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With GVHD (Graft Versus Host Disease)
Description: Acute grade 2 to 4 Graft versus host disease( GVHD )for patients who were able to be analyzed by measuring the T cell counts for increased CD3+ before and after lenalidomide.
Time Frame: Up to 6 months after allotransplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 21 | 8 | 9
Participants | 0 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study drug to 30 days post study drug completion (May 2009 to November 2015)
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 2/21 | 1/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/21 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 19/21 | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=21) | Group 2 (N=8) | Group 3 (N=9)
Skin GVHD (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
TIA (Blood and lymphatic system disorders) | 1 | 0 | 0
Graft Failure (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=21) | Group 2 (N=8) | Group 3 (N=9)
Epitaxis (Blood and lymphatic system disorders) | 1 | 0 | 0
Graf Failure (Blood and lymphatic system disorders) | 0 | 2 | 1
DVT (Cardiac disorders) | 4 | 0 | 1
A-fib (Cardiac disorders) | 1 | 0 | 1
Angina (Cardiac disorders) | 1 | 0 | 0
Hypertension (Cardiac disorders) | 3 | 1 | 0
Hypotension (Cardiac disorders) | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Ascites (Hepatobiliary disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 11 | 3 | 1
GI GVHD (Gastrointestinal disorders) | 14 | 1 | 6
Nausea (Gastrointestinal disorders) | 19 | 6 | 9
Elevated creatinine (Renal and urinary disorders) | 6 | 3 | 1
Cystitis (Renal and urinary disorders) | 5 | 0 | 1
Elevated Bilirubin (Hepatobiliary disorders) | 7 | 2 | 0
Liver GVHD (Hepatobiliary disorders) | 1 | 0 | 1
Transminitis (Hepatobiliary disorders) | 9 | 3 | 1
Nuetropenic infection (Infections and infestations) | 4 | 4 | 3
Infection (Infections and infestations) | 16 | 6 | 6
Hyperglycemia (Endocrine disorders) | 3 | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Occular GVHD (Eye disorders) | 3 | 2 | 1
Pnuemonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Skin GVHD (Skin and subcutaneous tissue disorders) | 11 | 5 | 7
Skin Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT00899431/Prot_SAP_000.pdf